CLINICAL TRIAL: NCT04166903
Title: Prospective Long Term Follow-up Analysis of Exercise-induced Physiological Changes in Male Runners
Brief Title: Prospective Follow-up, Marathon, Long Term, Inflammation and Cardiovascular System
Acronym: Pro-MagIC
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: Balgrist University Hospital (Other); Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Principal Investigator, Johannes Scherr, Prof. Dr. med. Johannes Scherr, Balgrist University Hospital
Other Study IDs: ProMagIC-Study
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2020-03

CONDITIONS: Participants of the Be-MaGIC-Study 2009
Keywords: Prolonged exercise, marathon, cardiovascular disease, long term
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample: whole blood, serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Pro-MagIC is a prospective observational study and includes participants of the Be-MaGIC-Study 2009 (n=277/NCT00933218). We aim to detect exercise-induced physiological changes (inter alia of the cardiovascular system) induced by repetitive ultra-endurance strain over a period of 10 years.

DETAILED DESCRIPTION:
Physical activity is associated with health benefits. Acute prolonged and strenuous exercise, i.e. Marathon running, leads to hemodynamic, endothelial and myocardial functional changes. Whether these myocardial, endothelial and hemodynamic changes can also develop and persist through repetitive extreme and prolonged physical activity is currently still a matter of controversy. In addition, it is not known whether adaptations and changes over time can develop into clinically relevant cardiovascular events with negative health consequences in healthy athletes. The aim of this study is to detect exercise-induced physiological changes (inter alia of the cardiovascular system) induced by repetitive ultra-endurance strain over a period of 10 years.

For this purpose, 277 male participants from the Be-MaGIC study (Marathon 2009) are examined in this prospective observational study. A single examination with the following components will take place: Anthropometry, clinical examination, laboratory, resting / exercise electrocardiography cardiopulmonary stress test, echocardiography, and fundus camera. Further examinations will be conducted in participants with abnormal examination results in line with current clinical recommendations.

ELIGIBILITY:
Inclusion Criteria:

Declaration of consent Participants must have participated in the Be-MaGIC study in 2009

* current age: 30 - 70 years
* sex: male

Exclusion Criteria:

-

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants of the Be-MaGIC-Study (2009)
Sampling Method: Non-Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Changes of right ventricular systolic function (RV-EF) | 10 years
  Echocardiography

SECONDARY OUTCOMES:
Changes in left ventricular ejection fraction (LV-EF) | 10 years
  Echocardiography
Changes in left ventricular diastolic function (E/e´) | 10 years
  Echocardiography
Change in cardiac markers (e.g. cardiac Troponin) | 10 years
  Clinical chemistry (blood samples)
Change in inflammation markers (e.g. C-reactive Protein) | 10 years
  Clinical chemistry (blood samples)
Change in microcirculation (e.g. arteriolar-to-venular ratio) | 10 years
  Static Retinal Vessel Analyzer
Change in macrocirculation (e.g. Intima media thickness) | 10 years
  Carotid sonography
Change of prevalence of cardiovascular diseases | 10 years
  Questionnaire
Association between changes of aforementioned parameters (see Topics 1-8) and potential underlying causes (e.g. sports history like number of ultraendurance competitions) in the examined cohort | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schindler, MD, Study Director — Department of Prevention, Rehabilitation and Sports Medicine, Munich, Germany; Johannes Scherr, MD, Principal Investigator — University Hospital Balgrist, University Zurich, Switzerland; Martin Halle, MD, Study Director — Department of Prevention, Rehabilitation and Sports Medicine, Munich, Germany
Locations (1):
- Department of Prevention, Rehabilitation and Sports Medicine, Munich, Germany, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matsushima M, Bryan GT. Early induction of mouse urinary bladder ornithine decarboxylase activity by rodent vesical carcinogens. Cancer Res. 1980 Jun;40(6):1897-901. PMID 7371022
- [Derived] Schoenfeld J, Schindler MJ, Haller B, Holdenrieder S, Nieman DC, Halle M, La Gerche A, Scherr J. Prospective long-term follow-up analysis of the cardiovascular system in marathon runners: study design of the Pro-MagIC study. BMJ Open Sport Exerc Med. 2020 Jul 19;6(1):e000786. doi: 10.1136/bmjsem-2020-000786. eCollection 2020. PMID 32704381